CLINICAL TRIAL: NCT04506320
Title: Novel Drugs (Immuno-modulating Agents, Protesome Inhibitors, Monoclonal Antibodies) After Allogeneic Transplant in Patients With Multiple Myeloma: an Observational Retrospective Study
Brief Title: Novel Drugs After Allo-HSCT in Patients With Multiple Myeloma
Acronym: NEW_ALL_MM
Status: Completed | Type: Observational
Sponsor: Gruppo Italiano Trapianto di Midollo Osseo (Other)
Collaborators: Azienda Ospedaliero-Universitaria Careggi (Other)
Responsible Party: Sponsor
Other Study IDs: GITMO-NEW_ALLO_MM
Record Dates: First submitted 2020-08-07; First posted 2020-08-10 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Multiple Myeloma; Stem Cell Transplant
Keywords: Allogeneic haematopoietic stem cell transplantation; Multiple Myeloma; Immuno-modulating agents; Protesome inhibitors; Monoclonal antibodies
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Multiple myeloma: Adult with diagnosis of multiple myeloma treated with Allo-HSCT from related - HLA identical or volunteer unrelated donor or haploidentical related donor performed from January 1, 2009 to december 31, 2018

SUMMARY:
This is a retrospective observational study of epidemiological surveillance, multicenter, non-profit, spontaneous, Italian on patients submitted to allo-HSCT among Italian Transplant Centers GITMO.

This study will evaluate all consecutive adult patients who received novel drugs after hematopoietic stem cell transplantation from related and unrelated donors between January 1, 2009 to December 31, 2018 in GITMO-affiliated Centers.

This study will evaluate approximately 300 subjects (with competitive enrolment) from GITMO investigational centers.

DETAILED DESCRIPTION:
This is a retrospective, observational multicenter, non-profit, spontaneous, Italian study organized under the auspices of the Gruppo Italiano Trapianti di Midollo Osseo that involves the principal Centers active in transplantation of any kind of hematopoietic stem cells in Italy.

Multiple myeloma is a neoplastic plasma cell disorder characterized by clonal proliferation of malignant plasma cells in the bone marrow and the presence of a monoclonal protein in the blood and/or urine, resulting in myeloma-defining events. The outcomes of patients with Multiple myeloma have improved significantly due to the introduction of novel agents; however, the disease remains incurable for most patients. Allogeneic hematopoietic stem cell transplantation has a curative potential by employing the donor immune system to eradicate malignant plasmacells, commonly referred to as the graft-versus-myeloma effect. However, despite this proven graft-versus-myeloma effect, the associated severe toxicity as treatment-related mortality mainly induced by myeloablative conditioning strategies and, above all, high relapse rate are important concerns and the place and role of allogeneic hematopoietic stem cell transplantation in Multiple myeloma remain challenging. In this regard, the International Myeloma Working Group together with the Blood and Marrow Transplant Clinical Trials Network, the American Society of Blood and Marrow Transplantation, and the European Society of Blood and Marrow Transplantation agreed that allogeneic hematopoietic stem cell transplantation should be considered an appropriate therapy for all eligible patients with early relapse (occurring within 24 months) after primary therapy that included the new proteasome inhibitors and immunomodulatory drugs and autologous stem cell transplantation and/or high-risk features.

allogeneic hematopoietic stem cell transplantation might represent an interesting platform for the use of rescue treatments based on novel drugs after the relapse. This observation might reflect the fact that allogeneic hematopoietic stem cell transplantation can modify the biology of the disease, directly targeting the myelomatous plasma cells as well as the microenvironment, and the well-documented graft-versus-myeloma effect induced by reactive allogeneic T cells may persist after relapse and contribute to an enhanced disease response. Novel agent-based combinations should be considered also in association with donor lymphocyte infusion. Monoclonal antibodies have emerged as the new option for treatment of patients with relapsed and refractory MM.

This scenario might represent a good opportunity to evaluate the efficacy of novel agents before and after transplantation.

The general objectives of this study are to retrospectively investigate the outcome of patients with Mieloma multiple after allogeneic hematopoietic stem cell transplantation and the first purpose of this study is to describe the overall survival at 2 years after allogeneic hematopoietic stem cell transplantation.

The secondary objectives are described Progression Free Survival, the incidence of acute and chronic graft versus host disease, describe the hematological and non-hematological toxicity of drugs administered after allogeneic hematopoietic stem cell transplantation and describe the Non-relapse- mortality.

Data will be stored using database Promise and specific e-CRFs. Data Center will perform extensive consistency checks and issue. Query Forms in case of inconsistent data. Follow-up period for the evaluation of survival will be from the date of transplant until 24 months post-transplant or death.

The study will be conducted according to the principles of Good Clinical Practice, the current Italian and European laws and regulations, in agreement with the declaration of Helsinki. The protocol has been written and the study will be conducted according to The International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use Harmonized Tripartite Guideline for Good Clinical Practice, issued by the European Union. The responsible Local Ethical Committee approval must be obtained before starting the trial. A copy of the patient informed consent form must be submitted to the appropriate authority or committee, together with the protocol for written approval. Written approval of the protocol and informed consent by the responsible and appropriate authority or committee must be obtained prior to recruitment of patients to the study.

ELIGIBILITY:
Inclusion Criteria Written and signed study informed consent Multiple myeloma Allogeneic transplantation from related - HLA identical Allogeneic transplantation from volunteer unrelated donor allogeneic transplantation from haploidentical related donor Myeloablative or reduced intensity conditioning regimen

Exclusion Criteria Second or further allogeneic transplant Plasma cell leukemia Non measurable disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Multiple Myeloma who had received novel drugs after allogeneic transplantation (allo-HSCT) from related and unrelated donor between January 1, 2009 to December 31, 2018.
  Each enrolled patient will have a two-year of follow-up from the allogeneic transplant date
Sampling Method: Probability Sample
Enrollment: 202 (Actual)
Dates: Start 2021-12-17 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Overall Survival (OS) | these outcome measures will be assessed at 2 year from transplant
  OS is defined as the time from transplant to the date of death due to any cause or to the last date the patient was known to be alive (censored observation) or to the date of the data cut-off for final analysis

SECONDARY OUTCOMES:
Progression Free Survival 1 (PFS1) | these outcome measures will be assessed at 2 year from transplant
  PFS1 is defined as the time interval from allo-HSCT until the first disease progression or death
Progression Free Survival 2 (PFS2) | These outcome measures will be assessed at 2 year from transplant
  PFS2 is defined as the time interval from allo-HSCT until the second disease progression or death, estimating the impact of both first- and second-line therapies on outcome.
Acute Graft-versus-Host Disease (aGVHD) | These outcome measures will be assessed at 100 days from transplant
  cumulative incidence of acute GvHD (grade II-IV)
Chronic Graft-versus-Host Disease (cGVHD) | These outcome measures will be assessed at 2 year from transplant
  Cumulative incidence and severity of chronic graft-versus-host disease
Non-Relapse Mortality (NRM) | These outcome measures will be assessed at 2 year from transplantation
  Cumulative incidence of Non-Relapse Mortality is defined as death due to any other cause than progression of malignancy after allogeneic stem cell transplantation.

CONTACTS AND LOCATIONS:
Overall Officials: Chiara Nozzoli, Principal Investigator — Azienda Ospedaliero-Universitaria Careggi
Locations (2):
- Italy (2):
  - Azienda Ospedaliera di Careggi, Florence
  - Clinica Ematologica - Policlinico Universitario, Udine

IPD SHARING:
Plan to Share IPD: No